CLINICAL TRIAL: NCT06421545
Title: Resilient Together for Dementia: A Live Video Resiliency Dyadic Intervention for Persons With Dementia and Their Care-partners Early After Diagnosis
Brief Title: Resilient Together for Dementia
Acronym: RT-D ADRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sarah Bannon, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GCO 23-0519; 1K23AG075188-01A1 (NIH)
Record Dates: First submitted 2024-04-30; First posted 2024-05-20 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer's Disease and Related Dementias
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Pilot RT-D Dyads (Experimental): Persons living with dementia (PWDs) and their spousal care-partners
  Interventions: Behavioral: Resilient Together for Dementia

INTERVENTIONS:
Behavioral: Resilient Together for Dementia — A novel live video dyadic resiliency intervention
  Other Names: RT-D

SUMMARY:
The proposed study will establish the feasibility, acceptability and credibility of a novel live video dyadic resiliency intervention, Resilient Together for Dementia (RT-D), aimed at preventing chronic emotional distress and preserving quality of life among dyads at risk for chronic emotional distress early after a diagnosis of Alzheimer's disease or a related dementia (ADRD).

DETAILED DESCRIPTION:
Both persons living with dementia (PWDs) and their spousal care-partners experience high levels of clinically elevated emotional distress, which can become chronic without treatment and negatively impact the health, quality of life, communication, and care-planning of both partners. A tailored dyadic intervention, such as the proposed Resilient Together for Dementia, delivered over live video to this at risk population during the window of opportunity when PWDs can participate has the potential to prevent chronic emotional distress and preserve quality of life for PWDs and their loved ones.

ELIGIBILITY:
PWD inclusion criteria are:

* Recent (~1 month) chart documented ADRD diagnosis,
* ADRD symptom onset after age 65 ,
* cognitive assessment scores and symptoms consistent with early stage dementia, as determined by the Clinical Dementia Rating Scale scores of .5 or 1.0
* cognitive awareness of his/her problems (as determined by the treating neurologist), and
* ability to understand study and research protocol, as determined by a standardized teach-back method assessment84.

Additional inclusion criteria for dyads are:

* English speaking adults (18 years or older),
* dyad lives together,
* at least one partner endorses clinically significant emotional distress during screening (>7 on Hospital Anxiety and Depression scale subscales)

Exclusion Criteria:

* patient is deemed inappropriate by the neurology team,
* either partner has a co-occurring terminal illness,
* patient was diagnosed with forms of dementia with clinical profiles that would preclude participation (e.g., Frontotemporal Dementia- behavioral variant), as determined by treatment team.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-04-19 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Proportion of potential eligible participants | After each dyad completion, throughout study of 1.5-2 months
  Feasibility of recruitment - Recruitment will be monitored by screening clinic visits for potentially eligible individuals and review recruitment progress in weekly meetings to promote completion within the study time frame. Recruitment will be monitored but will not set official benchmarks and modify procedures after each dyad.

SECONDARY OUTCOMES:
Proportion of participants screened | After each dyad completion, throughout study of 1.5-2 months
  Feasibility of screening - the portion of individuals who undergo screening that screen eligible and ineligible, and the reasons for ineligibility with detailed descriptions will be monitored and will review progress in weekly team meetings. Screening will be monitored but will not set official benchmarks and modify procedures after each dyad.
Proportion of participants who consent or not consent to participate | After each dyad completion, throughout study of 1.5-2 months
  Feasibility of consent by keeping a record of all individuals who complete screening that consent, refuse to consent, and the reasons for refusal will be monitored and will review progress in weekly team meetings. Feasibility of consent will be monitored but will not set official benchmarks and modify procedures after each dyad.
Proportion of sessions participants attend | After each dyad completion, throughout study of 1.5-2 months
  Feasibility of treatment -The number of sessions that enrolled dyads attend as well as missed sessions, treatment dropouts, and reasons for non attendance will be monitored and will review progress in weekly meetings. Feasibility of treatment will be monitored but will not set official benchmarks and modify procedures after each dyad.
Change in Hospital Anxiety and Depression Scale (HADS) | Baseline and 6 weeks (post-intervention)
  Change in emotional distress assessed with the Hospital Anxiety and Depression Anxiety Scale which is a 14-items scale with responses scored from 0-3, scores for each subscale (anxiety and depression) from 0 (normal) to 21 (severe symptoms). Scores for the entire scale is 0 to 42, with higher score indicating more distress.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Bannon, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Brain Injury Research Center at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data. Any purpose. Data are available indefinitely at (Link tbd).

REFERENCES:
- [Derived] Allison GO, McCage S, Brandt S, Presciutti M, Walker K, Cornelius T, Parker RA, Dams-O'Connor K, Dickerson B, Ritchie C, Vranceanu AM, Bannon SM. "We can do this. That I learned.": A nonrandomized open pilot of Resilient Together for Dementia, a post-diagnosis dyadic intervention. BMC Geriatr. 2026 Feb 12. doi: 10.1186/s12877-026-07059-9. Online ahead of print. PMID 41652334
- [Derived] McCage S, Walker K, Cornelius T, Parker RA, Dams-O'Connor K, Dickerson B, Ritchie C, Vranceanu AM, Bannon S. A Live Video Resiliency Dyadic Intervention for Persons With Dementia and Their Care-Partners Early After Diagnosis: Protocol for Open Pilot of Resilient Together for Dementia. JMIR Res Protoc. 2025 Jan 15;14:e60382. doi: 10.2196/60382. PMID 39814366

DOCUMENTS (1):
  • Informed Consent Form (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT06421545/ICF_000.pdf